CLINICAL TRIAL: NCT04578301
Title: Predicting Acute-on-Chronic Liver Failure After Surgical Intervention in Chronic Liver Disease
Acronym: PERSEVERE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Michael Praktiknjo, PI, University Hospital, Bonn
Other Study IDs: PERSEVERE
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Surgery; Acute-On-Chronic Liver Failure; Non-Cirrhotic Portal Hypertension
Keywords: ACLF; Acute-On-Chronic Liver Failure; Liver Cirrhosis; Portal Hypertension; Surgery; Non-Cirrhotic Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool and tissue samples from surgical specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery: Patients with and without liver cirrhosis undergoing surgery.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Prospective, observational study to define precipitants and predictors of development of Acute-on-Chronic Liver Failure (ACLF) after surgical interventions, allowing to develop a risk stratification for elective procedures in cirrhotic patients. As well as identifying molecular mechanisms of post-interventional ACLF and thus preparing the ground for development of new therapeutic approaches.

DETAILED DESCRIPTION:
Background: Acute-on-chronic liver failure (ACLF) is a recently discovered syndrome, which is understood as an acute deterioration of decompen-sated liver cirrhosis. It is defined on the basis of organ failure(s) and associated with high short-term mortality. ACLF is caused by a precipi-tating event that results in excessive systemic inflammation. ACLF is mostly precipitated and associated with bacterial infections but 40-50% of the underlying cause is unclear. Surgery, with or without liver involvement, has been defined as such a precipitating event. It is long known, that surgery in liver cirrhotic patients, depending on stage of cirrhosis as well as on type of surgery, bears a great risk but is still in-evitable in some cases. Child-Turquotte Score has been used for risk stratification of postoperative mortality. The development and out-come of ACLF after surgical interventions have not been characterized yet. In addition, underlying causes as well as molecular mechanism leading to ACLF after surgical intervention have not been identified. The aim of this trial is to further prospectively investigate patients with cirrhosis undergoing surgery to identify clinical markers and molecular mechanisms involved in development of ACLF.

Objectives: Defining precipitants and predictors of development of ACLF after surgical interventions, allowing to develop a risk stratification for elective procedures in cirrhotic patients.

Identifying molecular mechanisms of post-interventional ACLF and thus preparing the ground for development of new therapeutic approaches.

Study design: Prospective, observational study. Patients will be screened according inclusion/exclusion criteria. After informed consent sample processing will be possible from max. 1 week before scheduled surgery.

Primary endpoints: Development of ACLF within 28 and 90 days after visceral or non-visceral surgery in patients with portal hypertension (liver cirrhosis and idiopathic non-cirrhotic portal hypertension)

Secondary endpoints:

1. Mortality at 1 month, 3 months and 1 year.

   Following endpoints will be evaluated:

   " Time to death and mortality (overall and surgery-related) " Time to and rate of unplanned rehospitalizations after surgery " Any Infection and differentiated by site of infection (SBP, pneumonia, urinary tract infection, blood stream infection, Clostridium difficile-associated enterocolitis " Postsurgical acute hepatic decompensation and ACLF
2. To assess the changes in the intestinal microbiota in both groups and evaluate its effect on the primary endpoint.
3. To assess the potential socioeconomic impact.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult (≥18 years) patient
* With or without liver cirrhosis (diagnosed either histologically or by a combination of clinical, laboratory and radiological signs)
* Or Non-cirrhotic portal hypertension
* Non-pregnant, non-lactating females
* Ability to understand the patient information and to personally sign and date the informed consent to participate in the study
* The patient is co-operative and available for the entire study
* Provided written informed consent
* Indication for surgical intervention

Exclusion Criteria:

* Pregnant or lactating females
* Patients undergoing surgery as form of palliative cancer therapy
* Presence or history of severe extra-hepatic diseases
* HIV-positive patients
* Previous liver or other transplantation
* Patients with acute or subacute liver failure without underlying cirrhosis
* Patients who decline to participate
* Physician´s denial (e.g. the investigator considers that the patient will not follow the protocol scheduled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without liver cirrhosis and/or portal hypertension undergoing elective or emergency surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Episodes of Acute-on-Chronic Liver Failure (ACLF) | 90 days
  Development of ACLF after surgery

SECONDARY OUTCOMES:
1-year mortality | 12 months
  Death after surgery
Episodes of Acute Decompensation | 12 months
  Acute hepatic Decompensation after Surgery

OTHER OUTCOMES:
Intestinal Microbiota | 12 months
  Intestinal Microbiota will be assessed in stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Praktiknjo, MD, Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany